CLINICAL TRIAL: NCT03335969
Title: Evaluation of the HyGIeaCare Procedure for Patients With Chronic Constipation
Brief Title: HyGIeaCare Procedure for Chronic Constipation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients recruited
Sponsor: HyGIeaCare, Inc. (Industry)
Collaborators: Biostatistical Consulting, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGP-0003
Record Dates: First submitted 2017-10-30; First posted 2017-11-08 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-03

CONDITIONS: Constipation - Functional

STUDY DESIGN:
Intervention Model Description: Each patient will serve as their own control by comparing their bowel habits in a diary 4 weeks prior to colon irrigation to the bowel habits in their diary 4 weeks post colon irrigation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- pre colon irrigation diaries followed by post diaries (Experimental): 4 week bowel movement and rescue medication diaries will be compared to same diaries used 4 weeks after the colon irrigation procedure
  Interventions: Device: colon irrigation

INTERVENTIONS:
Device: colon irrigation — Study is to compare bowel movement patterns before and after colon irrigation.
  Other Names: HyGIeaCare System

SUMMARY:
To assess the safety and clinical effectiveness of using the FDA cleared HyGIeaCare System to relieve constipation in patients not responding to standard laxative treatment. Each patient will serve as their own control by comparing their bowel habits in a diary 4 weeks prior to colon irrigation to the bowel habits in their diary 4 weeks post colon irrigation.

DETAILED DESCRIPTION:
This study has a single center, prospective, open label design. Patients will serve as their own control.

The population will include patients with chronic constipation according to Rome III criteria who failed to improve with currently available therapy (osmotic and stimulant laxatives, used for at least one month at recommended dose).

Once patients are consented to participate in the study, they will complete the Gastrointestinal Symptom Severity Index (GISSI) questionnaire. Patients will complete the 4 Week Bowel Movement Diary and 4 Week Medication Use Diary for the 4-weeks prior to their HyGIeaCare procedure. The Medication Use Diary will include any rescue medications taken above and beyond what patients are taking as part of their constipation regimen.

The patient will schedule their HyGIeaCare procedure directly with the HyGIeaCare Clinic. The nurse manager can be reached at 480-750-2333. The clinic is located at 4001 E. Baseline Road, Gilbert, AZ. The nurse manager will provide the patient with any instructions needed prior to their HyGIeaCare procedure. HyGIeaCare will furnish the principle investigator with the complete patient care records after the irrigation procedure has been completed.

Following the 4 weeks post the patient's HyGIeaCare procedure, the patient will complete a new 4 Week Bowel Movement Diary and 4 Week Medication Use Diary for the 4-weeks post their HyGIeaCare procedure. The patient will bring these documents to their clinic follow-up visit. At this visit the patient will complete another GISSI questionnaire and will be evaluated for possible adverse events.

Patient data will be collected on hard copy case report forms (CRFs) and then entered into an electronic database.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has chronic constipation according to Rome III criteria
2. Patient has not experienced relief of symptoms following treatment with available therapies (osmotic and stimulant laxatives) for at least one month at recommended doses.

Exclusion Criteria:

1. Patient has functional bowel disorders characterized by alternating bowel habits (diarrhea/constipation)
2. Patient has secondary constipation (colonic obstruction, medications, metabolic cause)
3. Patient has any other condition that, in the opinion of the investigator, may adversely affect the compliance or safety of the patient or would limit the patient's ability to complete the study.
4. Patient has any of the contraindications listed below:

   1. Cardiac: Congestive heart failure (NYHA class III or IV or EF <50%)
   2. GI: Intestinal perforation, carcinoma of the rectum, fissures or fistula, severe hemorrhoids, abdominal hernia, recent colon or rectal surgery, or abdominal surgery
   3. GU: Renal insufficiency (CC < 60 ml/min/173m2), cirrhosis with ascites
   4. Abdominal surgery within the last 6 months
   5. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change in number of BMs | 8 weeks
  Change in the number of bowel movements per week from the baseline period (4 weeks) to the four weeks of the post-HyGIeaCare period.

SECONDARY OUTCOMES:
Change in constipation score and discomfort score (GISSI) | 8 weeks
  Gastrointestinal Symptom Severity Index (GISSI) constipation/difficult defecation cluster and abdominal pain/discomfort cluster
Change in rescue medications used | 8 weeks
  Review of the number of times rescue medications are used for constipation relief

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Umar, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

REFERENCES:
- [Background] Crowell MD, Umar SB, Lacy BE, Jones MP, DiBaise JK, Talley NJ. Multi-Dimensional Gastrointestinal Symptom Severity Index: Validation of a Brief GI Symptom Assessment Tool. Dig Dis Sci. 2015 Aug;60(8):2270-9. doi: 10.1007/s10620-015-3647-3. Epub 2015 Apr 5. PMID 25842355
- [Result] Sommers T, Corban C, Sengupta N, Jones M, Cheng V, Bollom A, Nurko S, Kelley J, Lembo A. Emergency department burden of constipation in the United States from 2006 to 2011. Am J Gastroenterol. 2015 Apr;110(4):572-9. doi: 10.1038/ajg.2015.64. Epub 2015 Mar 24. PMID 25803399
- See also: Randomized Trial Comparing High Volume Rectal Water Irrigation with Standard 4 L Split-Dose PEG Preparatoin before Colonoscopy — http://www.alliedacademies.org/articles/randomized-trial-comparing-high-volume-rectal-water-irrigation-with-standard-4-l-splitdose-peg-preparation-before-colonoscopy.pdf
- See also: Use of health care resources and cost of care for adults with constipation — https://www.google.com/search?q=Use+of+health+care+resources+and+cost+of+care+for+adults+with+constipation.+Clin+Gastroenterol+Hepatol.&rlz=1C1CHBF_enUS700US700&oq=Use+of+health+care+resources+and+cost+of+care+for+adults+with+constipation.+Clin+Gastroenterol+Hepatol.&aqs=chrome..69i57.814j0j4&sourceid=chrome&ie=UTF-8